CLINICAL TRIAL: NCT04339049
Title: Comparative Efficacy of Lidocaine Spray Versus Vaginal Misoprostol in Reducing Pain During IUD Insertion in Adolescents and Nulliparous Women: a Randomized Controlled Trial
Brief Title: Comparative Efficacy of Lidocaine Spray Versus Vaginal Misoprostol in IUD Insertion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Algazeerah hospital (Unknown)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lidocaine IUD
Record Dates: First submitted 2020-04-07; First posted 2020-04-08 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lidocaine spray (Experimental): four puffs (10 mg/puff) of lidocaine spray before tenaculum placement plus vaginal placebo 3 hours before IUD insertion
  Interventions: Drug: lidocaine spray
- vaginal misoprostol (Active Comparator): vaginal misoprostol 200 mcg given 3 hours before IUD insertion plus four puffs of saline spray before tenaculum placement
  Interventions: Drug: vaginal misoprostol
- placebo (Placebo Comparator): vaginal placebo given 3 hours before IUD insertion plus four puffs of saline spray before tenaculum placement
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lidocaine spray — four puffs (10 mg/puff) of lidocaine spray before tenaculum placement plus vaginal placebo 3 hours before IUD insertion
  Arms: lidocaine spray
Drug: vaginal misoprostol — vaginal misoprostol 200 mcg given 3 hours before IUD insertion plus four puffs of saline spray before tenaculum placement
  Arms: vaginal misoprostol
Drug: placebo — vaginal placebo given 3 hours before IUD insertion plus four puffs of saline spray before tenaculum placement
  Arms: placebo

SUMMARY:
the aim of the present study is to compare the safety and efficacy of lidocaine spray versus misoprostol in reducing pain during IUD insertion in adolescents and nulliparous women

ELIGIBILITY:
Inclusion Criteria:

* adolescent and young nulliparous women requesting IUD insertion

Exclusion Criteria:

* multiparous women, contraindications to IUD insertion or to study drugs

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
pain during IUD insertion | 5 minutes
  pain during IUD insertion evaluated by visual analog scale where 0 denotes no pain and 10 cm denotes the worst pain imaginable

SECONDARY OUTCOMES:
duration of IUD insertion | 5 minutes
  duration of IUD insertion from speculum in to speculum out

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Ashour, Giza, Egypt